CLINICAL TRIAL: NCT06734962
Title: Evaluation of Bone Regeneration After Apical Surgery Using Advanced Platelet-rich Fibrin: Utilization of Ultrasound for the Assessment of Periapical Lesions
Acronym: EBRAAPUU
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Riga Stradins University (Other)
Responsible Party: Principal Investigator, Aleksandra Karkle, Principal Investigator, Riga Stradins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-2/427/2021
Record Dates: First submitted 2024-12-05; First posted 2024-12-16 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Periapical Lesions
Keywords: Periapical healing; Apical Surgery; A-PRF; Ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Without A-PRF) (Other): During the surgery procedure A-PRF application is not intended.
  Interventions: Procedure: Apical surgery without using A-PRF
- Test group ( With A-PRF) (Experimental): During the surgery procedure A-PRF application is intended.
  Interventions: Procedure: Apical surgery procedure using A-PRF

INTERVENTIONS:
Procedure: Apical surgery procedure using A-PRF — Participants will undergo an apical surgery procedure using A-PRF. Before the surgery and at follow-ups, patients will undergo comprehensive evaluation using clinical, radiological, and ultrasonographic techniques.
  Arms: Test group ( With A-PRF)
Procedure: Apical surgery without using A-PRF — Participants will undergo an apical surgery procedure without using A-PRF. Patients will undergo comprehensive evaluation before the surgery and at follow-ups using clinical, radiological, and ultrasonographic techniques.
  Arms: Control group (Without A-PRF)

SUMMARY:
The study examines the impact of advanced platelet-rich fibrin (A-PRF) on bone regeneration in apical surgery compared to standard methods. It highlights the effectiveness of ultrasound as a diagnostic tool for assessing periapical lesions. Eligible participants were adults with specific periapical lesions following root canal treatment failures. Exclusions included patients outside specific criteria, like those with advanced periodontal disease or undergoing orthodontic treatment. Participants were randomized into two groups: one receiving A-PRF to enhance bone regeneration and a control group without it. Both groups underwent apical surgery under magnification, with different postoperative protocols. The study involved radiological and ultrasonographic evaluations of lesion size and bone healing at baseline, 6 months, and 12 months, alongside blood analyses for Vitamin D and cholesterol level to assess their potential impact on healing.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with precisely defined periapical lesions related to maxillary or mandibular incisors and premolar teeth as a sequel to persistent endodontic infection
2. Patients after root canal treatment/retreatment
3. Patients with or without the sinus tract
4. Patients with root perforations
5. Patients with clinical cases deemed unsuitable for non-surgical endodontic intervention
6. Patients with traumatic lesions clearly indicated for endodontic apical surgery.

Exclusion Criteria:

1. Patients younger than 18 years
2. Patients with lesions unrelated to the root apical area
3. Patients in possession of vital teeth with radiolucency in the apical region
4. Pregnant patients
5. Patients with non-restorable teeth
6. Patients with advanced periodontal disease
7. Patients with uncontrolled systemic health conditions
8. Patients receiving bisphosphonate therapy
9. Patients receiving orthodontic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-09-12 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Volumetric bone volume healing assessment | Baseline, 6 and 12 month
  Volumetric analysis of CBCT images will segment the defect in axial, sagittal, and coronal views. Bone volume will be measured in cubic millimeters (mm³) at pre-operative, 6-month, and 12-month follow-ups and compared between each other. Where 0 is - no periapical lesion/periapical lesion healed.

SECONDARY OUTCOMES:
Asessment of Ultrasound diagnostic accuracy for periapical lesion measurment | Baseline
  During the baseline assessment, the dimensions of periapical lesions will be measured in millimeters and using the classification:
  Category 1: no discernible periapical lesion was identified; Category 2: a periapical lesion was possibly present, however, the distinction was equivocal; Category 3: a periapical lesion was definitively observed. not unequivocal; Category 3: a periapical lesion was definitively observed. These measurements will then be analyzed in relation to images obtained through periapical radiography as well as those from cone beam computed tomography (CBCT). This comparison aims to evaluate the accuracy and reliability of different imaging techniques in assessing the size of periapical lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- Riga Stradins University Institute of Stomatology, Riga, Latvia

IPD SHARING:
Plan to Share IPD: Undecided